CLINICAL TRIAL: NCT05621018
Title: A Randomized Controlled Trial of "Maze Out": A Serious Game to Improve Self-efficacy, Mutual Understanding and Improved Family Functioning in People With Eating Disorders.
Brief Title: "Maze Out": A Serious Game to Improve Self-efficacy and Mutual Understanding in Eating Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Maze Out
Record Dates: First submitted 2022-11-02; First posted 2022-11-17 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Eating Disorders
Keywords: serious games; coproduction; bulimia nervosa; anorexia nervosa; mHealth
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa; Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Patients will be introduced to Maze Out in an information meeting with the investigators and will afterwards receive a link with the game and a username. Each patient has to choose a code to start playing the game. The code will not be available for the investigators.
  Interventions: Device: Maze Out
- Control group (Active Comparator): Patients will be introduced to Maze Out. 15 weeks later they will follow the same procedure as intervention group.
  Interventions: Device: Maze Out

INTERVENTIONS:
Device: Maze Out — Play for 15 weeks, at list once a week the serious game: Maze Out

SUMMARY:
Eating Disorders (EDs) are mental disorders with long recovery time and high mortality. Despite the importance and extensive research in the field, an effective treatment for EDs has yet to be found.

In co-production with ED patients, clinicians, and technology experts a Serious Game called "Maze out" was developed and initially evaluated through a feasibility study. Maze out is an innovative first player tool focusing on improving self-efficacy, mutual understanding, and family functioning in adults with EDs.

The game has been evaluated through a usability study. Study findings demonstrate that patients found Maze out easy to use, meaningful and fun.

The usability study was thus a first step in developing and testing an evidence-based intervention to be implemented in the treatment repertoire of adolescents and adults with EDs.

The present study is a Randomized Controlled Trial, whereby the investigators will explore the effectiveness of Maze out as an additional treatment to Treatment as Usual (TAU)

ELIGIBILITY:
Inclusion Criteria:

* All sexes aged 18+
* Diagnosis of anorexia nervosa, bulimia nervosa, other eating disorders and eating disorders unspecified (ICD-10 codes: F.50.0-F.50.9)
* Receiving treatment from one of psychiatry centers in the Mental Health Services of Region South Denmark, or in Endocrinology Services specialized in ED of Region South Denmark; or living in a mental health care institution in Region of Southern Denmark.

Exclusion Criteria:

• No Danish speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy | at baseline, 8 weeks and 15 weeks
  measured by a 5-item self-efficacy questionnaire (5-item SE_ED), is a 5-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life when having an Eating Disorder.Min.score: 0, max.score:40; higher score shows better outcome.

SECONDARY OUTCOMES:
perceived help received from staff | baseline and after 15 weeks
  measured by Brief INSPIRE: has one total score, ranging from 0 (low recovery support) to 100 (high recovery support).
feelings of ineffectiveness and self-image | baseline and after 15 weeks
  measured by Eating Disorders Inventory (EDI-3): consists of 91 items organized onto 12 primary scales, consisting of 3 eating-disorder-specific scales and 9 general psychological scales that are highly relevant to, but not specific to, eating disorders.This secondary outcome will focus in two domains: Inefectiveness and Interpersonal problems
interpersonal and intrapsychic interactions | baseline, 8 weeks, 15 weeks
  measured by Structural Analysis of Social Behavior Questionnaire (SAS-B) Designed to measure the patient's perceptions of self and others, based on trait x state x situational philosophy and Structural Analysis of Social Behavior.can be used to assess interpersonal and intrapsychic interactions in terms of three underlying dimensions: (a) focus (other, self, introject), (b) affiliation-hostility (love-hate), and (c) interdependence-independence (enmeshment-differentiation).
family function | baseline, 8 weeks, 15 weeks
  measured by Family APGAR (Adaptability, Partnership, Growth, Affection, and Resolve) Scores range from 0 to 10 with higher scores indicating better functionality.
mental health literacy | baseline, 15 weeks
  measured by MHLS (The Mental Health Literacy Scale), The Mental Health Literacy Scale (MHLS) is a 35 item questionnaire looking at the respondents understanding of mental health.Max score=160; Min score=35

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Mercedes Guala, Odense C, Denmark

REFERENCES:
- [Derived] Guala MM, Bikic A, Bul K, Clinton D, Mejdal A, Nielsen HN, Stoving RK, Nielsen AS. Maze-Out: A Serious Game to Enhance Treatment for Eating Disorders. A Randomized Controlled Trial. Int J Eat Disord. 2025 Aug;58(8):1558-1571. doi: 10.1002/eat.24458. Epub 2025 May 19. PMID 40384493
- [Derived] Guala MM, Bikic A, Bul K, Clinton D, Mejdal A, Nielsen HN, Stenager E, Sogaard Nielsen A. "Maze Out": a study protocol for a randomised controlled trial using a mix methods approach exploring the potential and examining the effectiveness of a serious game in the treatment of eating disorders. J Eat Disord. 2024 Mar 1;12(1):35. doi: 10.1186/s40337-024-00985-2. PMID 38429839

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-03-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT05621018/SAP_000.pdf